CLINICAL TRIAL: NCT01841827
Title: The Headache Inducing Effects of Cilostazol on Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-2-2013-033
Record Dates: First submitted 2013-04-20; First posted 2013-04-29 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Active Comparator): Capsule of Cilostazol 200 mg are taken orally on each study day
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator): A capsule of placebo containing starch are taken orally on each study day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol
  Other Names: Pletal
  Arms: Cilostazol
Drug: Placebo
  Arms: Placebo

SUMMARY:
We will use Cilostazol as a tool to investigate its headache inducing effects in migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine without aura according to the IHS criteria from 2004.
* Healthy besides migraine

Exclusion Criteria:

* Tension-type headache more than 3 days per month
* Other types of primary headaches
* Pregnancy
* History of vascular diseases or psychiatric diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The incidens of headache or migraine after adminstration of Cilostazol in migraine patients compared to placebo. | Outcome measure will be done within 3 month. Final data will be presented within 6 months
  Rectruitment of 14 patients will be done during April and May. Experiments will be carried out in May and June. Each experiment day takes 1½ hour. Data analysis will be done in June and July. Final data will be presented within 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center & Department of Neurology, Copenhagen, Glostrup, Denmark